CLINICAL TRIAL: NCT01653743
Title: Open-Label, Parallel-Group, Randomized, Multicenter Phase III Trial to Compare the Efficacy and Safety of a 250 mcg SC Dose of MSJ-0011 to a 5,000 IU IM Dose of Urinary Human Chorionic Gonadotropin in Inducing Ovulation in Japanese Women Diagnosed With Anovulation or Oligo-Ovulation Secondary to Hypothalamic-Pituitary Dysfunction or Polycystic Ovarian Syndrome, and Who Are Undergoing Ovulation Induction With Follitropin Alfa
Brief Title: Trial to Assess the Clinical Efficacy and Safety of MSJ-0011 in Inducing Ovulation in Anovulatory or Oligo-ovulatory Japanese Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., Japan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR701173_002
Record Dates: First submitted 2012-07-20; First posted 2012-07-31 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Anovulation; Oligo-ovulation; Hypothalamic-pituitary Dysfunction; Polycystic Ovarian Syndrome
Keywords: Japanese
MeSH Terms: conditions — Anovulation; Polycystic Ovary Syndrome | interventions — Chorionic Gonadotropin; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSJ-0011 (Experimental)
  Interventions: Drug: MSJ-0011; Drug: Follitropin alpha
- urinary hCG (Active Comparator)
  Interventions: Drug: urinary hCG (u-hCG); Drug: Follitropin alpha

INTERVENTIONS:
Drug: MSJ-0011 — Subjects who underwent ovarian stimulation with follitropin alfa according to a low-dose step-up protocol for maximum of 28 days will receive a single dose of 250 microgram (mcg) MSJ-0011 (choriogonadotropin alfa [recombinant human Chorionic Gonadotropin, r-hCG]) subcutaneously (SC) within 32 hours after the last dose of follitropin alfa administration unless dominant follicle reached a mean diameter of greater than or equal to (>=) 18 millimeter (mm); not more than 3 follicles each with a mean diameter of >=16 mm and serum Estradiol (E2) level within an acceptable range for the number of follicle present, and not more than 2,000 picogram per milliliter (pg/mL).
  Arms: MSJ-0011
Drug: urinary hCG (u-hCG) — Subjects who underwent ovarian stimulation with follitropin alfa according to a low-dose step-up protocol for maximum of 28 days will receive a single dose of 5,000 IU u-hCG intramuscularly dose within 32 hours after the last dose of follitropin alfa administration unless dominant follicle reached a mean diameter of >=18 mm; not more than 3 follicles each with a mean diameter of >=16 mm and serum E2 level within an acceptable range for the number of follicle present, and not more than 2,000 pg/mL.
  Arms: urinary hCG
Drug: Follitropin alpha — Low-dose step-up protocol involves starting dose of follitropin alfa as 75 International Units (IU) subcutaneously per day ,increments by 37.5 IU every 7 days (Day 8, 15, 28) will be done if no ovarian response will be observed for maximum of 28 days.

SUMMARY:
This is an open-label, parallel-group, randomized, multicenter Phase III trial to compare the efficacy and safety of a single 250 microgram (mcg) subcutaneous dose of MSJ-0011 to a single 5,000 international units (IU) intramuscular dose of urinary human chorionic gonadotropin (hCG) in inducing ovulation in Japanese women diagnosed with anovulation or oligo-ovulation. Ovulation induction therapy will be undertaken with follitropin alfa. The primary objective is to show that MSJ-0011 is non-inferior to urinary hCG, as assessed by the ovulation rate.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged between 20 to 39 years inclusive and wishing to conceive
* Body Mass Index (BMI) of 17.0 to 29.0 kilogram per square meter (kg/m^2) inclusive (value up to first decimal place)
* No clinically significant abnormalities in serum thyroid stimulating hormone (TSH), dehydroepiandrosterone sulfate (DHEA-S), 17-hydroxyProgesterone (17-OHP), prolactin (PRL) and follicle-stimulating hormone (FSH) levels in the early follicular phase
* Anovulation or oligo-ovulation
* Any one of the following: spontaneous menstruation (at least twice per year) or a positive response to progestin as evidenced by menstruation.
* Eligible for ovarian stimulation with gonadotropins (e.g. documented failure to ovulate or achieve pregnancy with anti-estrogenic therapy such as clomiphene citrate)
* Male partner with normal semen analysis, as defined by World Health Organization (WHO) standards, within 12 months prior to date of informed consent
* Normal cervical smear results (Papanicolaou [PAP] score less than or equal to [<=] II) taken within 12 months prior to date of informed consent; if not available a cervical smear will be performed as part of screening
* Full comprehension of the trial and voluntary consent obtained in writing prior to participation in this trial

Exclusion Criteria:

* Infertility involving gynecological factors other than anovulation or oligo-ovulation secondary to hypothalamic-pituitary dysfunction (Grade 1 Amenorrhea, Oligomenorrhea or Anovulatory Cycles) or polycystic ovarian syndrome (PCOS) and for whom ovulation induction (OI) therapy is contraindicated
* Subjects with known surgical/histological diagnosis of endometriosis greater than Stage II (American Fertility Society classification), or endometriosis requiring treatment
* Infertility secondary to amenorrhea of uterine cause
* Infertility secondary to primary or premature ovarian failure
* Infertility secondary to known adrenal or thyroid dysfunction, or hyperprolactinemia
* Failure of ovulation in 2 or more consecutive previous cycles with any gonadotropins
* Subjects in whom pregnancy is contraindicated, e.g. malformations of sexual organs or fibroid tumors of the uterus incompatible with pregnancy
* Extrauterine pregnancy in the previous 3 months
* History or presence of intracranial tumor (e.g. hypothalamic or pituitary tumor)
* Presence of or suspected gonadotropin- or estrogen-dependent malignancy (e.g. ovarian, uterine or mammary carcinoma)
* Untreated endometrial hyperplasia
* Abnormal hemorrhage of the reproductive tract of unknown origin
* History of severe ovarian hyper stimulation syndrome (OHSS) (Classification of OHSS Severity, Japan Reproductive/Endocrine Working Group)
* Clinically significant systemic disease (e.g. insulin-dependent diabetes, epilepsy, severe migraine, intermittent porphyria, hepatic, renal or cardiovascular disease, severe corticosteroid-dependent asthma)
* Participation in another clinical trial within 3 months prior to date of informed consent or simultaneous participation in another clinical trial
* Gonadotropin treatment within 2 months prior to date of informed consent
* Legal incapacity or limited legal capacity

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2012-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., Japan
Locations (6):
- Japan (6):
  - Hanabusa Women's Central Fertility Clinic, Hyōgo
  - Bashamichi Ladies Clinic, Kanagawa
  - Sophia Ladies Clinic, Kanagawa
  - Ivf Namba Clinic, Osaka
  - Ivf Osaka Clinic, Osaka
  - Department of Obstetrics and Gynecology, Saitama Medical University Hospital, Saitama

RESULTS

PARTICIPANT FLOW:
Groups:
- MSJ-0011: Subjects who underwent ovarian stimulation with follitropin alfa according to a low-dose step-up protocol (starting dose of follitropin alfa as 75 International Units (IU) subcutaneously per day ,increments by 37.5 IU every 7 days was done if no ovarian response was observed) for maximum of 28 days received a single dose of 250 microgram (mcg) MSJ-0011 subcutaneously (SC) within 32 hours after the last dose of follitropin alfa administration unless dominant follicle reached a mean diameter of greater than or equal to (>=) 18 millimeter (mm); not more than 3 follicles each with a mean diameter of >=16 mm and serum Estradiol (E2) level within an acceptable range for the number of follicle present, and not more than 2,000 picogram per milliliter (pg/mL).
- u-hCG: Subjects who underwent ovarian stimulation with follitropin alfa according to a low-dose step-up protocol (starting dose of follitropin alfa as 75 IIU subcutaneously per day ,increments by 37.5 IU every 7 days was done if no ovarian response was observed) for maximum of 28 days received a single dose of 5,000 IU u-hCG intramuscularly dose within 32 hours after the last dose of follitropin alfa administration unless dominant follicle reached a mean diameter of >=18 mm; not more than 3 follicles each with a mean diameter of >=16 mm and serum E2 level within an acceptable range for the number of follicle present, and not more than 2,000 pg/mL.
Period: Overall Study
Arm/Group | MSJ-0011 | u-hCG
Started | 54 | 27
Completed | 50 | 27
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Investigator discretion | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all the subjects who received investigational medicinal product ([IMP]; MSJ-0011 or u-hCG)
Groups:
- Urinary Human Chorionic Gonadotropin (u-hCG): Subjects who underwent ovarian stimulation with follitropin alfa according to a low-dose step-up protocol (starting dose of follitropin alfa as 75 IIU subcutaneously per day ,increments by 37.5 IU every 7 days was done if no ovarian response was observed) for maximum of 28 days received a single dose of 5,000 IU u-hCG intramuscularly dose within 32 hours after the last dose of follitropin alfa administration unless dominant follicle reached a mean diameter of >=18 mm; not more than 3 follicles each with a mean diameter of >=16 mm and serum E2 level within an acceptable range for the number of follicle present, and not more than 2,000 pg/mL.
- Total: Total of all reporting groups
Arm/Group | MSJ-0011 | Urinary Human Chorionic Gonadotropin (u-hCG) | Total
Number analyzed (Participants) | 54 | 27 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.61 (3.303) | 30.67 (3.603) | 31.96 (3.506)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 27 | 81
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Ovulation Mid-luteal Serum Progesterone (P4) Level of Greater Than or Equal (>=) 5 Nanogram Per Milliliter (ng/mL) or Clinical Pregnancy
Description: Ovulation was defined as mid-luteal serum progesterone level of >= 5 ng/mL or clinical pregnancy. Clinical pregnancy was defined as the presence of at least a fetal sac on transvaginal ultrasound (TVUS).
Time Frame: Mid-luteal phase progesterone assessed (Day 5 to 10) or clinical pregnancy (Day 35 to 42) post hCG treatment
Population: The modified intent to treat (Mod ITT) population was defined as all subjects randomized to IMP (MSJ-0011 or u-hCG) and who completed the primary efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MSJ-0011 | u-hCG
Number analyzed (Participants) | 54 | 27
percentage of subjects | 100 [93.4 to 100] | 100 [87.2 to 100]

2. Secondary Outcome: Percentage of Subjects With Ovulation Mid-Luteal Serum Progesterone (P4) Level of Greater Than or Equal (>=) 9.4 Nanogram Per Milliliter (ng/mL) or Clinical Pregnancy
Description: Ovulation was defined as mid-luteal serum progesterone level of >= 9.4 ng/mL or clinical pregnancy. Clinical pregnancy was defined as the presence of at least a fetal sac on TVUS.
Time Frame: Mid-luteal phase progesterone assessed (Day 5 to 10) or clinical pregnancy (Day 35 to 42) post hCG treatment
Population: The Mod ITT population was defined as all subjects randomized to IMP (MSJ-0011 or u-hCG) and who completed the primary efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MSJ-0011 | u-hCG
Number analyzed (Participants) | 54 | 27
percentage of subjects | 96.3 [87.3 to 99.5] | 88.9 [70.8 to 97.6]

3. Secondary Outcome: Mid-luteal Endometrial Thickness
Description: Endometrial thickness was measured using TVUS.
Time Frame: Day 5 to 7 post hCG treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | MSJ-0011 | u-hCG
Number analyzed (Participants) | 54 | 27
millimeter | 11.6 (2.64) | 12.4 (2.58)

4. Secondary Outcome: Percentage of Participants With Biochemical Pregnancy
Description: Percentage of subjects with biochemical pregnancy was assessed. Biochemical pregnancy was defined as any miscarriage without any evidence of a fetal sac on TVUS on the Day 35 to 42 post hCG treatment, but with a positive serum β-hCG pregnancy test on Day 15 to 20 post hCG treatment (Beta-hCG level greater than [>] 10 IU/Liter)
Time Frame: Day 35 to 42 post hCG treatment
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MSJ-0011 | u-hCG
Number analyzed (Participants) | 54 | 27
percentage of subjects | 3.7 [0.5 to 12.7] | 3.7 [0.1 to 19.0]

5. Secondary Outcome: Percentage of Participants With Clinical Pregnancy
Description: Percentage of subjects with clinical pregnancy was assessed. Clinical pregnancy was defined as the presence of at least a fetal sac on TVUS.
Time Frame: Day 35 to 42 post hCG treatment
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MSJ-0011 | u-hCG
Number analyzed (Participants) | 54 | 27
percentage of subjects | 29.6 [18.0 to 43.6] | 33.3 [16.5 to 54.0]

ADVERSE EVENTS:
Time Frame: From signing of the informed consent document until Day 28-31 (for subjects who had a negative serum β-hCG pregnancy test on Day 15-20), or up to the Day 35-42 post hCG treatment (for subjects who have a positive serum β-hCG pregnancy test on Day 15-20).
Arm/Group | MSJ-0011 | u-hCG
Serious Adverse Events (participants affected / at risk) | 1/54 | 0/27
Other Adverse Events (participants affected / at risk) | 32/54 | 11/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSJ-0011 (N=54) | u-hCG (N=27)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSJ-0011 (N=54) | u-hCG (N=27)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Injection site bruising (General disorders) | 1 | 0
Injection site erythema (General disorders) | 5 | 2
Injection site pain (General disorders) | 2 | 3
Injection site swelling (General disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 4 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 6 | 3
Ovarian enlargement (Reproductive system and breast disorders) | 1 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 7 | 4
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other